CLINICAL TRIAL: NCT05698407
Title: Effect of Dexmedetomidine Plus Ropivacaine Versus Sufentanil Plus Ropivacaine for Epidural Labor Analgesia on Neonatal Outcomes: a Pilot Randomized Trial
Brief Title: Dexmedetomidine-Ropivacine Versus Sufentanil-Ropivacaine for Epidural Labor Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, MD, PHD, Professor and Chairman, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-368
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related
Keywords: epidural labor analgesia; dexmedetomidine; neonatal outcomes
MeSH Terms: interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, pilot trial with two parallel-arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants, attending anesthesiologists and other health-care team members, and outcome assessors are blinded to the study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): loading dose of 0.45 microgram/ml dexmedetomidine plus 0.09% ropivacaine, maintenance dose of 0.36 microgram/ml dexmedetomidine plus 0.07% ropivacaine
  Interventions: Drug: Dexmedetomidine
- Sufentanil (Active Comparator): loading dose of 0.45 microgram/ml sufentanil plus 0.09% ropivacaine, maintenance dose of 0.36 microgram/ml sufentanil plus 0.07% ropivacaine
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Dexmedetomidine — loading dose of 0.45 microgram/ml dexmedetomidine plus 0.09% ropivacaine, maintenance dose of 0.36 microgram/ml dexmedetomidine plus 0.07% ropivacaine.
  Other Names: Dexmedetomidine-ropivacaine combination
  Arms: Dexmedetomidine
Drug: Sufentanil — loading dose of 0.45 microgram/ml sufentanil plus 0.09% ropivacaine, maintenance dose of 0.36 microgram/ml sufentanil plus 0.07% ropivacaine.
  Other Names: Sufentanil-ropivacaine combination
  Arms: Sufentanil

SUMMARY:
Sufentanil-ropivacaine combination is commonly used for epidural labor anesthesia, but is associated with some adverse events. Dexmedetomidine is a high selective alpha2-adrenoceptor agonist. Mounting evidences show that dexmedetomidine-ropivacaine combination can also be used effectively for epidural labor analgesia. This pilot trial is designed to compare the effect of dexmedetomidine-ropivacaine combination versus sufentanil-ropivacaine combination on neonatal outcomes when used for epidural labor analgesia, and to test the feasibility of a future large randomized trial.

DETAILED DESCRIPTION:
Sufentanil combined with ropivacaine is commonly used for epidural labor anesthesia. However, this combination is associated with some adverse events including increased risk of neonatal depression. Dexmedetomidine is a high selective alpha2-adrenoceptor agonist and possesses opioid-sparing and analgesic effects when used in combination with local anesthetics. Recently published data suggest that dexmedetomidine-ropivacaine combination can effectively relieve labor pain.

We suppose that, when compared with traditional sufentanil-ropivacaine combination, the dexmedetomidine-ropivacaine combination used for epidural labor analgesia may reduce sufentanil-related adverse neonatal outcomes. The purpose of this pilot trial is to compare the effect of dexmedetomidine-ropivacaine combination versus sufentanil-ropivacaine combination used for epidural labor analgesia on neonatal outcomes, and also to test the feasibility of a future large randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years;
2. Single term pregnancy with vertex presentation planning vaginal delivery;
3. Planning to receive epidural labor analgesia.

Exclusion Criteria:

1. Presence of contraindications to epidural analgesia, which includes: (1) History of infectious disease of the central nervous system (poliomyelitis, cerebrospinal meningitis, encephalitis, etc.); (2) History of spinal or intra-spinal disease (trauma or surgery of spinal column, intra-spinal canal mass, etc.); (3) Systemic infection (sepsis); (4) Skin or soft tissue infection at the site of epidural puncture; (5) Coagulopathy.
2. Existence of bradycardia (heart rate <60 bpm), hypotension (SBP <90 mmHg) or severe hypertension (SBP ≥180mmHg), uncontrolled systemic comorbidities (i.e., diabetes or hepatic, renal or cardiac disease), American Society of Anesthesiologists (ASA) physical status ≥3.
3. History of psychiatric disease or epilepsia.
4. Allergy to study agents.
5. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Composite neonatal morbidity | Up to 24 hours after birth
  Included any of the following: 1-min or 5-min Apgar score less than 7, umbilical cord arterial PH less than 7.1, requirement for immediate assisted ventilation, neonatal intensive care unit or neonatal ward admission within 24 hours after birth.

SECONDARY OUTCOMES:
Duration of labor | From the begining of the first stage of labor until delivery of the placenta, up to 20 hours
  Durations of the first, second, and third stages of labor
Delivery mode | At the time of delivery
  The mode of delivery includes spontaneous delivery, instrumental delivery, and Cesarean delivery.
Epidural infusion volume | From the begining of epidural analgesia until childbirth, up to 20 hours
  Total epidural infusion volume and epidural infusion volume per hour
Subjective sleep quality score at the first night after childbirth | Up to 24 hours after childbirth
  Numeric Rating Scale (NRS) score of subjective sleep quality
The depression score assessed by Edinburgh Postnatal Depression Scale (EPDS) | At 42 days after childbirth
  The depression will be assessed with the Edinburgh Postnatal Depression Scale (EPDS; score range 0-30, with higher score indicating more severe depression). The assessment will be conducted by a telephone interview. A score of EPDS ≥10 was set as the threshold of postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijin, Bejing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AI, McCarthy RJ, Toledo P, Jones MJ, White N, Wong CA. Epidural Labor Analgesia-Fentanyl Dose and Breastfeeding Success: A Randomized Clinical Trial. Anesthesiology. 2017 Oct;127(4):614-624. doi: 10.1097/ALN.0000000000001793. PMID 28926440
- [Background] Armstrong S, Fernando R. Side Effects and Efficacy of Neuraxial Opioids in Pregnant Patients at Delivery: A Comprehensive Review. Drug Saf. 2016 May;39(5):381-99. doi: 10.1007/s40264-015-0386-5. PMID 26832926
- [Background] Hussain N, Grzywacz VP, Ferreri CA, Atrey A, Banfield L, Shaparin N, Vydyanathan A. Investigating the Efficacy of Dexmedetomidine as an Adjuvant to Local Anesthesia in Brachial Plexus Block: A Systematic Review and Meta-Analysis of 18 Randomized Controlled Trials. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):184-196. doi: 10.1097/AAP.0000000000000564. PMID 28178091
- [Background] Hetta DF, Fares KM, Abedalmohsen AM, Abdel-Wahab AH, Elfadl GMA, Ali WN. Epidural dexmedetomidine infusion for perioperative analgesia in patients undergoing abdominal cancer surgery: randomized trial. J Pain Res. 2018 Oct 30;11:2675-2685. doi: 10.2147/JPR.S163975. eCollection 2018. PMID 30464585
- [Background] Qian M, Gao F, Liu J, Xu P. Dexmedetomidine versus fentanyl as adjuvants to ropivacaine for epidural anaesthesia: A systematic review and meta-analysis. Int J Clin Pract. 2021 May;75(5):e13772. doi: 10.1111/ijcp.13772. Epub 2020 Dec 20. PMID 33078536
- [Background] Zhang X, Wang D, Shi M, Luo Y. Efficacy and Safety of Dexmedetomidine as an Adjuvant in Epidural Analgesia and Anesthesia: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Clin Drug Investig. 2017 Apr;37(4):343-354. doi: 10.1007/s40261-016-0477-9. PMID 27812971
- [Background] Liu L, Drzymalski D, Xu W, Zhang W, Wang L, Xiao F. Dose dependent reduction in median effective concentration (EC50) of ropivacaine with adjuvant dexmedetomidine in labor epidural analgesia: An up-down sequential allocation study. J Clin Anesth. 2021 Feb;68:110115. doi: 10.1016/j.jclinane.2020.110115. Epub 2020 Nov 1. PMID 33142249
- [Derived] Jin KX, Deng CM, Ding T, Qu Y, Wang DX. Impact of dexmedetomidine-ropivacaine versus sufentanil-ropivacaine combination for epidural labour analgesia on neonatal outcomes: a pilot randomised clinical trial. BMJ Open. 2024 Dec 22;14(12):e090208. doi: 10.1136/bmjopen-2024-090208. PMID 39806707